CLINICAL TRIAL: NCT06756152
Title: Prospective Pilot Study of the Clinical Efficacy and Safety of the Method for Preventing a Graft-versus-host Disease Through the Agency of Using the Combination of Post-transplantation Cyclophosphamide with Abatacept, Vedolizumab and Ruxolitinib At Children and Young Adults with Hemoblastosis After Hematopoietic Stem Cell Transplantation from an Unrelated or Haploidentic Donor
Brief Title: Preventing of GVHD with Post-transplantation Cyclophosphamide, Abatacept, Vedolizumab and Ruxolitinib At Children and Young Adults with Hemoblastosis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCHPOI-2024-10
Record Dates: First submitted 2024-12-13; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Biphenotypic Acute Leukemia; Acute Lymphoblastic Leukemia; Myeloblastic Leukemia; Bilinear Leukemia; Malignant Lymphoma, Non-Hodgkin; Myelodysplastic Syndrome
Keywords: Hematopoetic stem cell transplantation; posttransplant cyclophosphamide; vedolizumab; hematoblastosis; ALL; AML
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelomonocytic, Acute; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes | interventions — Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention of GVHD: Cyclophosphamide, Abatacept, Vedolizumab, Ruxolitinib (Experimental): GVHD prevention using a combination of post-transplantation cyclophosphamide in combination with abatacept, vedolizumab and Ruxolitinib in children and young adults with hematoloblastosis after myeloablative conditioning regimen
  Interventions: Drug: Conditioning regimen: Treosulfan 42 g/m2/course or total body irradiation 12 Gray/course, Etoposide 60 mg/kg , Fludarabine 150

INTERVENTIONS:
Drug: Conditioning regimen: Treosulfan 42 g/m2/course or total body irradiation 12 Gray/course, Etoposide 60 mg/kg , Fludarabine 150 — The most significant adverse events limiting the use of HSCT from an unrelated donor are graft-versus-host disease (GVHD) and prolonged immunodeficiency associated with the development of severe infectious complications. The use of post-transplant cyclophosphamide for the prevention of GVHD during allogeneic HSCT from unrelated and haploidentical donors has reduced the incidence of acute clinically significant GVHD in children to 25%, chronic GVHD to 12-30%, but the issue of GVHD control still remains extremely relevant. Emerging data on the use of abatacept, a selective blocker of the costimulatory signal from an antigen-presenting cell, in the prevention of intestinal GVHD and data on the effectiveness of Janus-kinase type 1/2 inhibitors (JAK-1/2) in the treatment and prevention of acute GVHD allow us to justify the use of these drugs in combination with post-transplant cyclophosphamide as a promising pharmacological platform for the prevention of GVHD.

SUMMARY:
GVHD prevention using a combination of post-transplantation cyclophosphamide in combination with abatacept, vedolizumab and Ruxolitinib in children and young adults with hematoloblastosis after myeloablative conditioning regimen with treosulfan/TBI, etoposide, fludarabine after HSCT from matched unrelated and haploidentical donors

DETAILED DESCRIPTION:
Conditioning regimen:

Treosulfan 42 g/m2/course on the days -5, -4, -3 or total body irradiation 12 Gray/course on the days -8, -7, -6 Etoposide 60 mg/kg on the days -6, -5. or Thiotepa 10 mg/kg -6,-5 Fludarabine 150 mg/m2/course on the days -6, -5, -4, -3, -2

Prevention of GVHD:

Cyclophosphamide 80 mg/kg/course on the days +3, +4 Abatacept 10 mg/kg/day on the days +5, +14, +28, +60, +90 Vedolizumab 10 mg/kg/day, max. 300 mg on the days 0, +14, +28, +60

Ruxolitinib 10 mg/m2 per os, from day -3 to day +90 (after HSCT), orally, twice a day.

Donor selection criteria

In case of detection of two or more suitable donors, the choice is made in favor of:

* CMV Compliance
* Sex of donor and recipient
* medical and psychological suitability and desire of the donor
* Compatibility by blood type

Duration of therapy

* 120 days (for patients with high risk of recurrence: positive minimal residual disease before HSCT, non-remission status after HSCT, patients diagnosed with juvenile myelomonocytic leukemia)
* 180 days (for the rest) Time of observation
* follow up during 3 years after HSCT

Criteria for premature stopping of the study

1. The probability of developing acute GVHD II-IV is above 40%, of which III-IV - above 15%
2. The probability of 100-day transplant-associated mortality is higher than 20%. Goal Evaluation Date Intermediate analysis after 1 year from the beginning. The final analysis is scheduled to take place 100 days after the last patient is included.

Data Monitoring and Management

1. Plan of initial examination of the patient

After signing the informed consent and registration, the patient undergoes an examination in accordance with the standard plan of pre-transplantation examination and additional examinations, including:

* Confirmation of remission status, determination of MRD, chimerism according to the protocol 1. Monitoring of donor chimerism in patients with acute leukemia Point Days Lines

  1 +30 day general, CD34
* Only if a relapse of the disease is suspected, cm can be sent to study chimerism:

  * General
  * Chimerism in the sorted MRD fraction 2. Minimal residual disease (MRD) monitoring in patients with ALL +30, +100 days after HSCT - for all patients: MRD (immunophenotyping), Cytogenetics (if it presence)

    + 60, +180 days after HSCT - for patients with MRD + or refractory before HSCT: MRD (immunophenotyping), Cytogenetics (if it presence) 3. Minimal residual disease (MRD) monitoring in patients with AML

    +100 days after HSCT - for all patients: MRD (immunophenotyping), Cytogenetics (if it presence)

    + 30, +180 days after HSCT - for patients with MRD + or refractory before HSCT: MRD (immunophenotyping), Cytogenetics (if it presence)

    4. Biobanking (KM, blood)

In this protocol, in addition to routine post-transplantation monitoring, the following studies are carried out:

• Study of the subpopulation composition of peripheral blood lymphocytes: B-cells: CD19

T-cells:

CD3/4/8/ TCR/gd CD3/4/8/45RA/CCR7 (CD197) CD3/4/31/45RA CD4/25/127

NK-compartment:

CD3/CD56

TCR repertoire:

Analysis multiplicity: +30, +60, +100, +180, +360 day The amount of blood for analysis is 5 ml in a test tube with EDTA.

* Pathogen-specific immunoreconstitution research - ELISPOT method for evaluating the production of gamma-interferon by peripheral blood mononuclears after incubation with microbial antigens. The main antigens studied are (CMV pp65, EBV, Adenovirus (AdvHexon), BK virus) Multiplicity of analysis of recipients: +30, +60, +100, +180, +360. The amount of blood for analysis on +30 days is 10 ml, subsequently - 5 ml in a test tube with EDTA.
* Virological monitoring by PCR weekly:

Blood: CMV, EBV, ADV by PCR method Chair: ADV MONITORING by PCR is carried out up to 100 days after CGSC. The exception is patients with viremia, or receiving immunosuppressive therapy on day 100.

in case of suspected visceral lesion: cerebrospinal fluid / bal / stool / urine / biopsy / other material

* Biobanking Multiplicity: + 30, +60, +100, +180, +360 Blood in a test tube with EDTA, used 2. Toxicity monitoring:
* Diagnosis and therapy of acute GVHD Clinical diagnosis and staging of acute GVHD is carried out in accordance with standard criteria (Appendix No. 3).

When an isolated rash appears, a skin biopsy is mandatory. When a clinic of acute GVHD appears with damage to the upper and lower gastrointestinal tract (nausea, vomiting, enterocolitis), gastroscopy with a biopsy of the gastric mucosa and colonoscopy with a floor biopsy is reokended.

The biopsy material should also be sent for virological examination. Before starting therapy, a consultation is held with the head of the protocol / appointed expert.

• Criteria for prescribing systemic immunosuppressive therapy: Acute GVHD stage I - therapy is not carried out Acute GVHF stage II-IV - methylprednisolone 1-2 mg / kg / day IV The period for assessing the response to first-line therapy: 72 hours, 7 days, 14 days from the start of therapy.

• Criteria for prescribing second-line therapy: progression of manifestations of O.RTPH after 72 hours or no improvement after 7 days or incomplete resolution of clinical and laboratory manifestations after 14 days

• Diagnosis and therapy of chronic GVHD: Diagnosis and staging of chronic GVHD are performed in accordance with THE NIH criteria (Appendix No. 4). Due to the fact that the development of chronic GVHD is one of the main parameters for the evaluation of the study, the diagnosis and staging of chronic GVHD are performed prospectively, monthly from the day +100, using a structured examination in accordance with Appendix No. 2.

Therapy of chronic GVHD is carried out in accordance with the standard adopted in the clinic

ELIGIBILITY:
Inclusion Criteria:

1. Patients under the age of 21 years with following diseases:

* acute lymphoblastic,
* myeloblastic,
* biphenotypic,
* bilinear leukemia,
* malignant lymphoma,
* myelodysplastic syndrome,

Exclusion Criteria:

Age over 21 years

* Patients with ALL outside clinical and hematological remission
* Clinical status:

  * Lansky/Karnowski index <70% (supplement No.1)
  * Heart function: left ventricular ejection fraction <40% according to ultrasound of the heart1
  * Kidney function: clearance of endogenous creatinine < 70 ml / min
  * Liver function: total bilirubin, ALT, AST, ALP > 2 norms
  * Lung function: lung capacity <50%, for children who cannot carry out of respiratory function - oxygen saturation during pulse oximetry <92%
* Uncontrolled viral, fungal or bacterial infection.
* Mental illness of the patient or caregivers, making it impossible to realize the essence of the study and compromising compliance with medical appointments and sanitary and hygienic regime 1 These patients may receive treatment according to the protocol, but the results will be evaluated separately

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
1. Cumulative Incidence stage II-IV after HSCT | up to 100 days
  Estimate the probability of developing acute GVHD stage II-IV after HSCT-
Kaplan Meier overal survival | up to 100 days
  Explore the safety based on an assessment of the frequency of occurrence severe (3-5 degrees) side effects of conditioning- 100-day transplant-associated mortality
1. Cumulative Incidence stage II-IV after HSCT | up to 100-day
  Estimate the probability of developing acute GVHD stage II-IV after HSCT
Kaplan Meier event free survival | during 1 month
  Explore the safety based on an assessment of the frequency of occurrence severe (3-5 degrees) side effects of conditioning
Kaplan Meier event free survival | up to 100 days
  Explore the safety based on an assessment of the frequency of occurrence severe (3-5 degrees) side effects of conditioning- 100-day transplant-associated mortality

SECONDARY OUTCOMES:
event-free survival | up to 100 days
  Probability of developing a relapse of the primary disease, transplantation-associated mortality on the horizon of 100 days, general and event-free survival
Cumulative Incidence of leukocyte engraftment | up to 30 days
  Probability and kinetics of engraftment of leukocyte and platelet sprouts of donor origin
Cumulative Incidence of platelet engraftment | up to 30 days
  Probability and kinetics of engraftment of leukocyte and platelet sprouts of donor origin
Cumulative Incidence reactivation of CMV | up to 6 mouth or up to immunreconstitution
  Probability of reactivation of CMV, EBV, AdV, HHV6 infection
box plot | up to 1 year
  Kinetics of general and pathogen-specific immunoreconstitution
Cumulative Incidence of chronic GVHD | up to 1 year
  Probability of the development of chronic GVHD, its severity and the nature of the involvement of organs and tissues.
Cumulative Incidence reactivation of EBV | up to 6 mouth or up to immunreconstitution
  Probability of reactivation of CMV, EBV, AdV, HHV6 infection
Cumulative Incidence reactivation of AdV | up to 6 mouth or up to immunreconstitution
  Probability of reactivation of CMV, EBV, AdV, HHV6 infection
Cumulative Incidence reactivation of HHV6 | up to 6 mouth or up to immunreconstitution
  Probability of reactivation of CMV, EBV, AdV, HHV6 infection

CONTACTS AND LOCATIONS:
Locations (1):
- National medical research center of pediatric haematology, oncology and immulogy named after Dmytriy Rogachyov, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided